CLINICAL TRIAL: NCT04472793
Title: Repeated Employee Testing for Understanding Our Recovery to Normal
Acronym: RETURN
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: RETURN
Record Dates: First submitted 2020-06-03; First posted 2020-07-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and DNA Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Full-Time CCHMC Employees
  Interventions: Diagnostic Test: SARS-CoV-2

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 — 1. Testing weekly samples from nasal swabs to promptly diagnose acute COVID-19 infection.
  2. Testing monthly serum samples to document post-viral infection.

SUMMARY:
The purpose of this research study is 1) to conduct a prospective longitudinal surveillance research trial, enrolling up to 200 CCHMC employees as they come back to work, and then following their clinical and laboratory parameters for up to 12 months; and 2) to support the ongoing development of diagnostic techniques for COVID-19. The overall goal is to investigate patterns of SARS-COV-2 infection, including immunological recovery and genetic risk factors, among CCHMC employees to better understand how to safely reintroduce the CCHMC work force back into their normal routines.

DETAILED DESCRIPTION:
As the global and pandemic spread of the novel coronavirus (SARS-CoV-2, COVID-19) continues, many knowledge gaps remain with regard to the epidemiology and transmission of infection, as well as the normal immunological responses after viral exposure. Cincinnati only recently (March 14, 2020) had its first confirmed case of COVID-19, and through shelter-in-place and social distancing efforts, has avoided the community spread experienced by some other large metropolitan areas. As investigators contemplate the gradual reintroduction of the Cincinnati Children's Hospital Medical Center (CCHMC) workforce back into the hospital, it is imperative that investigators determine the current prevalence of infection among CCHMC employees, measure the cumulative incidence of infection over the next 12 months, investigate the normal antibody patterns after infection, and help elucidate what constitutes a protective immunological response. Investigators have a unique but time-limited opportunity to optimally track the epidemiology and natural history of SARS-CoV-2 infection at CCHMC, including risk factors for transmission and immunological recovery. RETURN will investigate epidemiological and immunological features of SARS-CoV-2 virus infection in a limited cohort of CCHMC employees, as they return from the current shelter-at-home directive toward a normal work environment. By collecting and analyzing weekly serial samples for SARS-CoV-2 (nasal swab for virus by PCR) and monthly serological exposure (serum antibodies by ELISA), investigators will determine the prevalence and cumulative incidence of exposure to SARS-CoV-2; document the antibody responses over time; identify cases of apparent viral recrudescence or re-infection; and create models of transmission risk among CCHMC employees.

ELIGIBILITY:
Inclusion Criteria:

* Current full-time employees at Cincinnati Children's Hospital
* Age: >18.0 years of age, at the time of enrollment
* Cell phone that can be used for text messaging or web-based viewing of surveys
* Willing and able to provide informed consent
* Ability to comply with all study related evaluations and follow-up

Exclusion Criteria:

* Previous proven SARS-CoV-2 infection (positive PCR-based molecular test)
* Any condition or illness that makes study participation ill-advised
* Currently or planning to enroll in a COVID-19 vaccine or prophylaxis study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult men and women who are employed full time at Cincinnati Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The 6-month cumulative incidence of acquired COVID infection in the study cohort. | Weekly for 6 months
  Acquired COVID is defined as testing negative for COVID at baseline and having 1 or more weekly nasal swab samples testing positive for the virus by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Russell Ware, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Mary Allen Staat, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No